CLINICAL TRIAL: NCT06639321
Title: The Safety and Efficacy of the Percutaneous Left Ventricular Assist System Versus ECMO for Intraoperative Circulatory Support During High-risk Percutaneous Coronary Intervention (PCI): a Prospective, Multi-center, Randomized Controlled Study
Brief Title: Phimume® Percutaneous Left Ventricular Assist System Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai NewMed Medical Co., Ltd. (Industry)
Collaborators: Shanghai Phigine Medical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Phimume -2024
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Ventricular Assist System; high-risk PCI
MeSH Terms: conditions — Coronary Artery Disease | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- percutaneous left ventricular assist system (Experimental): Subjects with coronary artery disease receiving high-risk PCI will be supported by Percutaneous Ventricular Assist System during the procedure.
  Interventions: Device: Percutaneous Ventricular Assist System
- extracorporeal membrane oxygenation (ECMO) (Active Comparator): Subjects with coronary artery disease receiving high-risk PCI will be supported by ECMO during the procedure.
  Interventions: Device: extracorporeal membrane oxygenation (ECMO)

INTERVENTIONS:
Device: Percutaneous Ventricular Assist System — Percutaneous Ventricular Assist System provides intraoperative circulatory support during high-risk PCI.
  Arms: percutaneous left ventricular assist system
Device: extracorporeal membrane oxygenation (ECMO) — ECMO provides intraoperative circulatory support during high-risk PCI.
  Arms: extracorporeal membrane oxygenation (ECMO)

SUMMARY:
The primary purpose of this clinical trial is to evaluate the safety and efficacy of the percutaneous left ventricular assist system versus extracorporeal membrane oxygenation (ECMO) for circulatory support during high-risk PCI.

DETAILED DESCRIPTION:
This prospective, multi-center, randomized controlled clinical trial of the Percutaneous Ventricular Assist System is designed to measure the incidence of freedom from major adverse cardiovascular and cerebrovascular events (MACCE) at 30 days after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old≤ patient age ≤90 years old AND patient is not in pregnancy or lactation;
2. Patients who have been evaluated by two or more cardiovascular surgeons as unsuitable for conventional surgery; or patients who have refused conventional surgery after adequate communication from the surgeon and who are at high risk for conventional surgery;
3. Left Ventricular Ejection Fraction (LVEF) ≤ 35% AND at least one of the following criteria:

   * Intervention on the last patent coronary conduit, or
   * Intervention on an unprotected left main coronary artery Or b) LVEF ≤ 30% and intervention in patient presenting with triple vessel disease.
4. Patient who can understand the purpose of the trial and volunteer to participate in, sign the informed consent form and are willing to accept relevant examinations and clinical follow-ups.

Exclusion Criteria:

1. Pre-procedure cardiac arrest within 24 hours of enrolment requiring CPR;
2. Pre-procedure ST-segment myocardial infarction within 24 hours of enrolment;
3. Patient is in cardiogenic shock;
4. Mural thrombus in the left ventricle;
5. Post-infarction ventricular septal rupture, or atrial septal or ventricular septal defects;
6. The presence of mechanical aortic or mitral valve or heart constrictive device;
7. The presence of aortic stenosis (aortic orifice area ≤1.5cm²)；
8. The presence of moderate to severe aortic or mitral or tricuspid insufficiency;
9. The presence of severe peripheral vascular disease that would preclude the placement of the percutaneous mechanical circulatory assist device;
10. Severe aortic diseases such as aortic dissection and aortic aneurysm;
11. Active infective endocarditis or other active infections;
12. Chronic renal insufficiency (creatinine clearance≤30ml/min);
13. Liver dysfunction (elevation of liver enzymes and bilirubin levels to ≥3xULN or INR≥2);
14. The presence of uncorrectable abnormal coagulation (platelet count≤75,000/mm^3 or INR≥2.0 or fibrinogen≤1.50 g/l);
15. The presence of uncorrected moderate to severe anemia (hemoglobin <90 g/L);
16. History of stroke or TIA within 1 month of enrolment;
17. Allergy or intolerance to contrast media, anticoagulant and antiplatelet drugs (e.g., bivalirudin, low molecular heparin, aspirin, clopidogrel, Ticagrelor, etc.);
18. Severe pulmonary artery hypertension (pulmonary artery systolic pressure >70 mmHg);
19. Participation in clinical trials of other drugs or medical devices prior to enrollment that have not yet reached the primary outcome of research;
20. Patient with poor compliance and could not complete the study as required determined by the investigator.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-14 (Estimated); Primary Completion 2025-11-14 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of freedom from major adverse cardiovascular and cerebrovascular events (MACCE) | 30 days after procedure
  MACCE defined as death, myocardial infarction, stroke, and target vessel revascularization.

SECONDARY OUTCOMES:
Incidence of death | 30 days, 90 days after procedure
  Rate of all-cause death during the trial.
Incidence of myocardial infarction | 30 days, 90 days after procedure
  Rate of patients with myocardial infarction during the trial.
Incidence of stroke | 30 days, 90 days after procedure
  Rate of patients with stroke during the trial.
Incidence of target vessel revascularization | 30 days, 90 days after procedure
  Rate of patients with target vessel revascularization during the trial.
Incidence of need for cardiac operation or thoracic or abdominal vascular operation or vascular operation for limb ischemia | 30 days, 90 days after procedure
  Rate of patients with unplanned cardiac operation or thoracic or abdominal vascular operation or vascular operation for limb ischemia during the trial.
Incidence of acute kidney injury Remove | 30 days, 90 days after procedure
  Rate of patients with acute kidney injury during the trial.
Incidence of cardiopulmonary resuscitation or ventricular arrhythmia requiring cardioversion | 30 days, 90 days after procedure
  Rate of patients with cardiopulmonary resuscitation or ventricular arrhythmia requiring cardioversion during the trial.
Incidence of increasing in aortic insufficiency by more than one grade | 30 days, 90 days after procedure
  Rate of patients with increasing in aortic insufficiency by more than one grade during the trial.
Incidence of severe hypotension | 30 days, 90 days after procedure
  Rate of patients with severe hypotension during the trial. Severe hypotension defined as systolic blood pressure or augmented diastolic pressure (whichever is greater) <90 mmHg for ≥5 min requiring inotropic/pressor medications or IV fluid.
Incidence of freedom from major adverse cardiovascular and cerebrovascular events (MACCE) | 90 days after procedure
  Rate of patients with freedom from major adverse cardiovascular and cerebrovascular events (MACCE) during the trial. MACCE defined as death, myocardial infarction, stroke, and target vessel revascularization.
Hemodynamic support success rate during PCI procedure | During procedure
  Hemodynamic support success is defined as (1) Percutaneous mechanical circulatory assist device was delivered and activated successfully, and withdrawn from the body successfully; (2) Hemodynamic stability during procedure (defined as mean arterial pressure (MAP) <60mmHg for no more than 10 minutes during the PCI procedure and additional pressor medication is not required).
Technical success rate | mmediately after procedure
  Technical success is defined as (1) Hemodynamic support success; (2) Coronary revascularization success (defined as ①residual stenosis <30% after coronary stent implantation; ②restoration of TIMI anterograde flow of II or III).
Procedural success rate | Immediately after procedure
  Procedure success is defined as (1) Technical success; (2) Freedom from serious in-hospital procedural complications
Change in LVEF compared to baseline | 30 days, 90 days after procedure
  LVEF is assessed at 30 days, 90 days after procedure, and compared to baseline
Improvement in cardiac function | 30 days, 90 days after procedure
  Cardiac function is evaluated based on NYHA classification and compared to baseline. New York Heart Association (NYHA) Functional Classification includes four categories(CLASS I to CLASS IV, higher class mean a worse outcome) based on physical activity limitations.
Evaluation of Experimental device performance | Immediately after procedure
  Performance evaluation includes the catheter pump and extracorporeal control device (For each assessment: 1-10 points；1=worst, 5=moderate, 10=best).

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Study Chair — The General Hospital of Northern Theater Command
Locations (6):
- China (6):
  - The Second Hospital of Jilin University, Jilin, Changchun
  - West China Hospital, Sichuan University, Chengdu, Chengdu
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - General Hospital of Northern Theater Command, Shenyang, Liaoning